CLINICAL TRIAL: NCT04290559
Title: Long-term Monitoring After Persistent Atrial Fibrillation Ablation and Correlation to Quality of Life
Brief Title: Persistent Atrial Fibrillation Ablation and Correlation to Quality of Life
Acronym: LEARN-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Newmarket Electrophysiology Research Group Inc (Other)
Responsible Party: Sponsor
Other Study IDs: NERG-04
Record Dates: First submitted 2020-02-11; First posted 2020-03-02 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation
Keywords: Catheter ablation; Quality of life; Atrial fibrillation burden; Persistent atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Reveal LINQ ILR implant before AF ablation — Patients will undergo insertion of a LINQ ILR before the atrial fibrillation ablation performed according to standard clinical practice.

SUMMARY:
The primary objective of this study is to determine the atrial fibrillation burden reduction, or absolute atrial fibrillation burden, associated with improvement in quality of life in patients undergoing ablation of persistent atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is associated with a higher risk of stroke, heart failure and deterioration in patients' quality of life and it also has great effect on health care resource utilization due to increasing morbidity and mortality. Catheter ablation has shown to improve patients' quality of life (QOL), even in those who undergo a repeat procedure, equalizing healthy population and lowering subsequent health care resource utilization.

Success rates are usually based on an endpoint of total elimination of AF, typically absence of any AF recurrence >30 seconds. While this is a high standard for clinical trial reporting, it does not necessarily measure the "clinical" success, since many patients will experience significant reduction in their AF burden with accompanying improvement in their functional status despite having ongoing brief recurrences of AF.

This is a prospective non-randomized, single-arm, cohort study. 200 patients with persistent atrial fibrillation undergoing catheter ablation will be enroled. AF burden post procedure will be evaluated with continuous monitoring with an implantable loop recorder (ILR) to assess recurrences and AF burden. QOL will be measured using the CCS-SAF severity scale, SF-36 and AFEQT scales pre-ablation and at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients undergoing first-time or redo AF ablation.
* Persistent or long-standing persistent AF
* Symptomatic atrial fibrillation
* Willing and able to provide informed consent.
* Willing and able to set up and utilize MyCareLink® home monitor and be remotely monitored
* Atrial fibrillation burden equal or more than 80% prior to the ablation

Exclusion Criteria:

* Paroxysmal AF
* If the patient has had a cardioversion within 2 months of the ablation
* Patients with contraindication to oral or intravenous anticoagulation.
* Contraindication to implantation of an ILR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent or long-standing persistent atrial fibrillation and an AF burden of equal or more than 80%, referred for an atrial fibrillation catheter ablation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
AF burden correlated with change in QOL. | 12 months, 24 months
  AF burden change and absolute AF burden correlated with change in QOL mesured at 12 and 24 months after the AF ablation

SECONDARY OUTCOMES:
Freedom of atrial arrhythmia | 12 months, 24 months
  Freedom of atrial tachycardia/atrial flutter/atrial fibrillation (> 30 sec) at 12 and 24 months after the ablation
Economic evaluation | 12 months, 24 months
  Change in AF burden correlated with change of health care resource utilization
Incidence of silent AF recurrences | 12 months, 24 months
  Total asymptomatic AF burden (Percent time in AF)
Impact of antiarrhythmic treatment | 12 months
  Compare quality of life on and off antiarrhythmic medications using 36-Item Short Form Survey (SF-36) scale: range 0-100, 100 is best.

CONTACTS AND LOCATIONS:
Locations (1):
- Southlake Regional Health Centre, Newmarket, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No